CLINICAL TRIAL: NCT03449134
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 12-Month Study to Evaluate the Efficacy and Safety of MK-7264 in Adult Participants With Chronic Cough (PN027)
Brief Title: A Study of Gefapixant (MK-7264) in Adult Participants With Chronic Cough (MK-7264-027)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-027; MK-7264-027 (Other: Merck Protocol Number); 2017-000537-31 (EudraCT Number); 184098 (Registry Identifier: JAPAN-CTI)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Intervention Model Description: Participants with refractory or unexplained chronic cough will be randomized to 1 of 3 treatment groups during the Treatment Period: Placebo, gefapixant 15 mg twice daily (BID), or gefapixant 45 mg BID. Participants will remain on their assigned treatment throughout the study. A safety follow-up phone call will be conducted at a minimum of 14 days after last dose of study treatment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants receive dose-matched placebo tablets twice daily (BID) during the 12-week main study period and 40-week extension period.
  Interventions: Drug: Placebo
- Gefapixant 15 mg BID (Experimental): Participants receive a gefapixant 15 mg tablet and placebo tablet to match gefapixant 45 mg BID during the 12-week main study period and 40-week extension period.
  Interventions: Drug: Placebo; Drug: Gefapixant
- Gefapixant 45 mg BID (Experimental): Participants receive a gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the 12-week main study period and 40-week extension period.
  Interventions: Drug: Placebo; Drug: Gefapixant

INTERVENTIONS:
Drug: Placebo — Participants receive dose-matched placebo tablets orally BID during the 12-week main study period and during the 40-week extension period.
Drug: Gefapixant — Gefapixant 15 mg or 45 mg tablet administered orally BID during the 12-week main study period and during the 40-week extension period, according to randomization.
  Other Names: MK-7264
  Arms: Gefapixant 15 mg BID; Gefapixant 45 mg BID

SUMMARY:
The main objectives of this study will be to evaluate the efficacy of gefapixant in reducing cough frequency as measured over a 24-hour period at Week 12, and to evaluate the safety and tolerability of gefapixant. The primary hypothesis is that at least one gefapixant dose is superior to placebo in reducing coughs per hour (over 24 hours) at Week 12.

DETAILED DESCRIPTION:
The study will include a screening period to determine participant inclusion, and the Baseline visit will include 24 hours of objective measurement of cough. The study will consist of two treatment periods, a main 12-week treatment period and a 40-week extension period (52 weeks total treatment), followed by a 14-day telephone follow-up period.

Participants at selected sites and countries who complete the main and extension study periods may consent to participate in an observational, 3-month, Off-treatment Durability Study Period, which extends the Estimated Study Completion Date. The Off-treatment Durability Study Period will explore the impact of withdrawing gefapixant in refractory or unexplained chronic cough participants who have been treated for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography scan of the thorax (within 5 years of Screening/Visit 1 and after the onset of chronic cough) not demonstrating any abnormality considered to be significantly contributing to the chronic cough or any other clinically significant lung disease in the opinion of the principal investigator or the sub-investigator
* Has had chronic cough for at least 1 year with a diagnosis of refractory chronic cough or unexplained chronic cough
* Female participants are eligible if not pregnant, not breastfeeding, and either not of childbearing potential, or agree to follow contraceptive guidance
* Provides written informed consent and is willing and able to comply with the study protocol (including use of the digital cough recording device and completion of study questionnaires)

Exclusion Criteria:

* Is a current smoker or has given up smoking within 12 months of Screening
* Has forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC) ratio <60%
* Has a history of respiratory tract infection or recent clinically significant change in pulmonary status
* Has a history of chronic bronchitis
* Is currently taking an angiotensin converting enzyme inhibitor (ACEI), or has used an ACEI within 3 months of Screening
* Has an estimated glomerular filtration rate (eGFR) <30mL/min/1.73 m^2 at Screening OR eGFR ≥30 mL/min/1.73 m^2 and <50 mL/min/1.73 m^2 at Screening with unstable renal function
* Has a history of malignancy <=5 years
* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence
* Has a history of anaphylaxis or cutaneous adverse drug reaction (with or without systemic symptoms) to sulfonamide antibiotics or other sulfonamide-containing drugs
* Has systolic blood pressure >160 mm Hg or diastolic blood pressure >90 mm Hg at Screening
* Has a known allergy/sensitivity or contraindication to gefapixant
* Has donated or lost >=1 unit of blood within 8 weeks prior to the first dose of gefapixant
* Has previously received gefapixant or is currently participating in or has participated in an interventional clinical study
* Had significantly abnormal laboratory tests at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (156):
- United States (27):
  - Research Solutions of Arizona PC ( Site 0036), Litchfield Park, Arizona
  - Medical Research of AZ ( Site 0060), Scottsdale, Arizona
  - Biosolutions Clinical Research Center ( Site 0070), La Mesa, California
  - Center for Clinical Trials, LLC ( Site 0059), Paramount, California
  - Sher Allergy Specialists/Center For Cough ( Site 0078), Largo, Florida
  - Well Pharma Medical Research, Corp. ( Site 0093), Miami, Florida
  - Florida Pulmonary Research Institute, LLC ( Site 0019), Winter Park, Florida
  - Midwest Allergy Sinus Asthma, SC ( Site 0081), Normal, Illinois
  - Cotton-O'Neil Clinical Research Center ( Site 0052), Topeka, Kansas
  - BreatheAmerica Inc ( Site 0048), Shreveport, Louisiana
  - Clinical Research Institute LLC ( Site 0004), Minneapolis, Minnesota
  - The Center for Pharmaceutical Research PC ( Site 0016), Kansas City, Missouri
  - American Health Research ( Site 0082), Charlotte, North Carolina
  - Clinical Research of Gastonia ( Site 0043), Gastonia, North Carolina
  - Bernstein Clinical Research Center, LLC ( Site 0005), Cincinnati, Ohio
  - Vital Prospects Clinical Research Institute, PC ( Site 0037), Tulsa, Oklahoma
  - Asthma Nasal Disease & Allergy Research Center of New England ( Site 0075), East Providence, Rhode Island
  - Sirius Clinical Research, LLC ( Site 0102), Austin, Texas
  - Pharmaceutical Research & Consulting, Inc. ( Site 0029), Dallas, Texas
  - Mainland Medical Research Institute ( Site 0003), Dickinson, Texas
  - Diagnostics Research Group ( Site 0035), San Antonio, Texas
  - Allergy & Asthma Center ( Site 0001), Waco, Texas
  - Intermountain Clinical Research ( Site 0033), Draper, Utah
  - Charlottesville Medical Research Center, LLC ( Site 0006), Charlottesville, Virginia
  - Pulmonary Associates of Richmond Inc. ( Site 0101), Richmond, Virginia
  - National Clinical Research-Richmond, Inc. ( Site 0073), Richmond, Virginia
  - Lung and Sleep Specialists ( Site 0091), Williamsburg, Virginia
- Argentina (9):
  - InAER Investigaciones en Alergia y Enfermedades Respiratorias ( Site 0324), Caba, Buenos Aires
  - Fundacion CIDEA ( Site 0323), Ciudad de Buenos Aires, Buenos Aires
  - Instituto Ave Pulmo ( Site 0322), Mar del Plata, Buenos Aires
  - Centro Medico Privado de Reumatologia ( Site 0309), San Miguel de Tucumán, Tucumán Province
  - Investigaciones en Patologias Respiratorias ( Site 0325), San Miguel de Tucumán, Tucumán Province
  - CEMEDIC - Centro de Especialidades Medicas ( Site 0304), Buenos Aires
  - Centro Medico Dra De Salvo ( Site 0310), Buenos Aires
  - Hospital Privado Universitario de Cordoba ( Site 0313), Córdoba
  - Fundacion Scherbovsky ( Site 0300), Mendoza
- Canada (7):
  - Canadian Phase Onward Inc. ( Site 0509), Toronto, Ontario
  - Recherche GCP Research ( Site 0500), Montreal, Quebec
  - 167877 Canada Inc. Dr. Jaime Del Carpio ( Site 0506), Montreal, Quebec
  - Dynamik Research ( Site 0505), Pointe-Claire, Quebec
  - Diex Recherche Quebec Inc ( Site 0515), Québec, Quebec
  - Q & T Research Sherbrooke Inc. ( Site 0512), Sherbrooke, Quebec
  - CIC Mauricie Inc. ( Site 0503), Trois-Rivières, Quebec
- Czechia (4):
  - MUDr. I. Cierna Peterova s.r.o. ( Site 0707), Brandýs nad Labem
  - Plicni ambulance ( Site 0701), Rokycany
  - Plicni stredisko Teplice s. r. o ( Site 0700), Teplice
  - Pneumologie Varnsdorf S.R.O. ( Site 0706), Varnsdorf
- Denmark (3):
  - CCBR AS Aalborg, Center for Clinical & Basic Research ( Site 0802), Aalborg
  - Herlev Hospital ( Site 0803), Herlev
  - CCBR AS Vejle, Center for Clinical & Basic Research ( Site 0801), Vejle
- France (5):
  - Hopital Cavale Blanche ( Site 0909), Brest
  - Hopital Nord du Marseille ( Site 0910), Marseille
  - Hopital Arnaud de Villeneuve ( Site 0905), Montpellier
  - CHU Hotel Dieu Nantes ( Site 0906), Nantes
  - CHU de Toulouse - Hopital Larrey ( Site 0900), Toulouse
- Hungary (5):
  - Dr Kenessey Albert Korhaz-Rendelointezet ( Site 1200), Balassagyarmat
  - Erzsebet Gondozohaz ( Site 1207), Gödöllő
  - Petz Aladar Megyei Oktato Korhaz ( Site 1206), Győr
  - Synexus Magyarorszag Kft. ( Site 1210), Gyula
  - CRU Hungary KFT ( Site 1205), Miskolc
- Israel (5):
  - Hillel Yaffe Medical Center ( Site 1303), Hadera
  - Carmel Medical Center ( Site 1305), Haifa
  - Meir Medical Center ( Site 1301), Kfar Saba
  - Rabin Medical Center ( Site 1302), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 1304), Ramat Gan
- Japan (38):
  - National Hospital Organization Nagoya Medical Center ( Site 1539), Nagoya, Aichi-ken
  - Nagoya City University Hospital ( Site 1528), Nagoya, Aichi-ken
  - National Hospital Organization Ehime Medical Center ( Site 1556), Tōon, Ehime
  - Idaimae Minamiyojo Int Clinic ( Site 1521), Sapporo, Hokkaido
  - Terada Clinic Respiratory Medicine & General Practice ( Site 1565), Himeji, Hyōgo
  - Kinki Central Hospital ( Site 1576), Itami, Hyōgo
  - Itami City Hospital ( Site 1580), Itami, Hyōgo
  - National Hospital Organization Ibarakihigashi National Hospital ( Site 1526), Naka-gun, Ibaraki
  - Ishikawa Prefectural Central Hospital ( Site 1554), Kanazawa, Ishikawa-ken
  - Kanazawa University Hospital ( Site 1536), Kanazawa, Ishikawa-ken
  - Komatsu Municipal Hospital ( Site 1508), Komatsu, Ishikawa-ken
  - Kamei Internal Medicine and Respiratory Clinic ( Site 1509), Takamatsu, Kagawa-ken
  - Fujisawa City Hospital ( Site 1505), Fujisawa, Kanagawa
  - Yokohama City Minato Red Cross Hospital ( Site 1506), Yokohama, Kanagawa
  - Medical Corporation Shintokai Yokohama Minoru Clinic ( Site 1568), Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital ( Site 1533), Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center ( Site 1503), Yokohama, Kanagawa
  - Matsusaka City Hospital ( Site 1525), Matsusaka, Mie-ken
  - Nagaoka Red Cross Hospital ( Site 1507), Nagaoka, Niigata
  - National Hospital Organization Minami-Okayama Medical Center ( Site 1553), Tsukubo-gun, Okayama-ken
  - Urasoe General Hospital ( Site 1572), Urasoe, Okinawa
  - Osaka Habikino Medical Center ( Site 1546), Habikino, Osaka
  - Kawaguchi Respiratory Clinic ( Site 1504), Higashiosaka, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 1519), Sakai, Osaka
  - Tokyo Medical University Hachioji Medical Center ( Site 1569), Hachiōji, Tokyo
  - National Hospital Organization Tokyo National Hospital ( Site 1557), Kiyose, Tokyo
  - National Hospital Organization Disaster Medical Center ( Site 1558), Tachikawa, Tokyo
  - Shimonoseki City Hospital ( Site 1573), Shimonoseki, Yamaguchi
  - National Hospital Organization Fukuoka Hospital ( Site 1552), Fukuoka
  - Hiroshima Allergy & Respiratory Clinic ( Site 1529), Hiroshima
  - Kyoto University Hospital ( Site 1547), Kyoto
  - JA Niigatakoseiren Niigata Medical Center ( Site 1522), Niigata
  - Shizuoka Prefectural Hospital Organization Shizuoka General Hospital ( Site 1524), Shizuoka
  - Juntendo University Hospital ( Site 1578), Tokyo
  - Tokyo Shinagawa Hospital ( Site 1560), Tokyo
  - Showa University Hospital ( Site 1531), Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 1574), Tokyo
  - Tokyo Metropolitan Geriatric Hospital ( Site 1577), Tokyo
- Peru (4):
  - Clinica Ricardo Palma ( Site 1802), San Isidro, Lima region
  - Hospital Nacional Adolfo Guevara Velasco ( Site 1808), Cusco
  - Asociacion Civil por la Salud ( Site 1805), Lima
  - Hospital Chancay y Servicios Basicos de Salud ( Site 1810), Lima
- Poland (9):
  - Prywatny Gabinet Internistyczno ( Site 1928), Bialystok
  - Centrum Medycyny Oddechowej Mroz Spolka Jawna ( Site 1918), Bialystok
  - Centrum Medyczne Pratia Bydgoszcz ( Site 1418), Bydgoszcz
  - Centrum Medyczne Pratia Czestochowa ( Site 1926), Częstochowa
  - Centrum Medyczne Pratia Gdynia ( Site 1910), Gdynia
  - Specjalistyczny osrodek .All-Med. Grazyna Pulka ( Site 1919), Krakow
  - USK nr 1 ( Site 1921), Lodz
  - Prywatny Gabinet Specjalistyczny ( Site 1927), Lodz
  - NZOZCentrum Medyczne Kermed ( Site 1905), Żnin
- South Korea (12):
  - Wonju Severance Christian Hospital ( Site 2214), Wŏnju, Gangwon-do
  - Hallym University Sacred Heart Hospital ( Site 2208), Anyang-si, Gyeonggi-do
  - Ajou University Hospital ( Site 2211), Suwon, Gyeonggi-do
  - Incheon St. Mary s Hospital ( Site 2200), Incheon
  - Seoul National University Hospital ( Site 2210), Seoul
  - The Catholic University of Korea Eunpyeong St Mary s Hospital ( Site 2209), Seoul
  - Severance Hospital ( Site 2204), Seoul
  - Konkuk University Medical Center ( Site 2205), Seoul
  - Asan Medical Center ( Site 2203), Seoul
  - Samsung Medical Center ( Site 2212), Seoul
  - The Catholic University of Korea St. Mary s Hospital ( Site 2215), Seoul
  - Korea University Guro Hospital ( Site 2213), Seoul
- Spain (4):
  - Hospital Clinic ( Site 2302), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 2309), Madrid
  - Hospital Parc Tauli ( Site 2308), Sabadell
  - Hospital Clinico Universitario de Santiago ( Site 2303), Santiago de Compostela
- Taiwan (5):
  - Changhua Christian Hospital ( Site 2403), Changhua
  - Chang Gung Medical Foundation - Keelung Branch ( Site 2404), Keelung
  - Far Eastern Memorial Hospital ( Site 2402), New Taipei City
  - Taichung Veterans General Hospital ( Site 2401), Taichung
  - National Taiwan University Hospital ( Site 2400), Taipei
- Turkey (Türkiye) (6):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2613), Ankara
  - I.U. Cerrahpasa Tip Fakultesi Gogus Hastaliklari Anabilim Dali ( Site 2600), Fatih
  - Yedikule Gogus Hast. ve Gogus Cer. Egitim ve Arastirma Hastanesi ( Site 2601), Istanbul
  - Kocaeli Universitesi Tip Fakultesi ( Site 2611), Kocaeli
  - Recep Tayyip Erdogan Universitesi Tip Fakultesi Egitim ve Aras. Has ( Site 2620), Rize
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi ( Site 2606), Samsun
- Ukraine (3):
  - F.G.Yanovskyy Institute of Phthisiology and Pulmonology ( Site 2830), Kyiv
  - City Polyclinic N20 ( Site 2822), Odesa
  - Private Small-Scale Enterprise Medical Centre "Pulse" ( Site 2815), Vinnytsia
- United Kingdom (10):
  - Royal Preston Hospital ( Site 2709), Preston, Lancashire
  - Medinova Lakeside Dedicated Research Centre ( Site 2710), Corby, Northamptonshire
  - Belfast City Hospital ( Site 2705), Belfast
  - Broomfield Hospital ( Site 2722), Chelmsford
  - Glenfield Hospital ( Site 2701), Leicester
  - Royal Brompton Hospital ( Site 2703), London
  - Wythenshawe Hospital ( Site 2700), Manchester
  - Churchill Hospital ( Site 2706), Oxford
  - Rothwell Medical Centre ( Site 2712), Rothwell
  - MeDiNova Yorkshire Dedicated Research Centre ( Site 2708), Shipley

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Dicpinigaitis PV, Birring SS, Blaiss M, McGarvey LP, Morice AH, Pavord ID, Satia I, Smith JA, La Rosa C, Li Q, Nguyen AM, Schelfhout J, Tzontcheva A, Muccino D. Demographic, clinical, and patient-reported outcome data from 2 global, phase 3 trials of chronic cough. Ann Allergy Asthma Immunol. 2023 Jan;130(1):60-66. doi: 10.1016/j.anai.2022.05.003. Epub 2022 May 13. PMID 35569802
- [Derived] McGarvey LP, Birring SS, Morice AH, Dicpinigaitis PV, Pavord ID, Schelfhout J, Nguyen AM, Li Q, Tzontcheva A, Iskold B, Green SA, Rosa C, Muccino DR, Smith JA; COUGH-1 and COUGH-2 Investigators. Efficacy and safety of gefapixant, a P2X3 receptor antagonist, in refractory chronic cough and unexplained chronic cough (COUGH-1 and COUGH-2): results from two double-blind, randomised, parallel-group, placebo-controlled, phase 3 trials. Lancet. 2022 Mar 5;399(10328):909-923. doi: 10.1016/S0140-6736(21)02348-5. PMID 35248186

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 732 participants randomized to the 52-week treatment period, 730 participants received at least 1 dose of study intervention. After the main study, 41 participants continued in an optional Off-Treatment observational study period (no treatment).
Groups:
- Placebo: Participants received dose-matched placebo tablets twice daily (BID) during the 12-week main study period and 40-week extension period.
- Gefapixant 15 mg BID: Participants received a gefapixant 15 mg tablet and placebo tablet to match gefapixant 45 mg BID during the 12-week main study period and 40-week extension period.
- Gefapixant 45 mg BID: Participants received a gefapixant 45 mg tablet and placebo tablet to match gefapixant 15 mg BID during the 12-week main study period and 40-week extension period.
Period: 52-Week Treatment Period
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Started | 244 | 244 | 244
Treated | 243 | 244 | 243
Completed | 199 | 200 | 184
Not Completed | 45 | 44 | 60
Not completed — Death | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Physician Decision | 2 | 3 | 3
Not completed — Screen Failure | 1 | 0 | 1
Not completed — Withdrawal by Subject | 37 | 39 | 55
Not completed — Site Closure | 1 | 0 | 0
Period: 12-Week Off-Treatment Durability Period
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Started | 10 (Not all participants continued in the optional Off-Treatment Period.) | 18 (Not all participants continued in the optional Off-Treatment Period.) | 13 (Not all participants continued in the optional Off-Treatment Period.)
Completed | 10 | 18 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID | Total
Number analyzed (Participants) | 244 | 244 | 244 | 732
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (13.1) | 59.6 (11.7) | 59.5 (13.1) | 59.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 181 | 181 | 544
  Male | 62 | 63 | 63 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 35 | 33 | 101
  Not Hispanic or Latino | 204 | 205 | 208 | 617
  Unknown or Not Reported | 7 | 4 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 8 | 21
  Asian | 35 | 35 | 34 | 104
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 4 | 11
  White | 190 | 195 | 187 | 572
  More than one race | 8 | 5 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Geographic Region [Count of Participants; unit: Participants] — Geographic region of enrollment with 5 categories: Asia-Pacific, Europe, North America, Others, and Missing.
  Participants
    Asia Pacific | 35 | 34 | 34 | 103
    Europe | 121 | 123 | 122 | 366
    North America | 56 | 55 | 56 | 167
    Others | 31 | 32 | 32 | 95
    Missing | 1 | 0 | 0 | 1
Baseline 24-hour Coughs per Hour [Mean (Standard Deviation); unit: coughs/hour] — 24-hour objective coughs per hour was defined as the total number of cough events during the monitoring period (24-hour interval) divided by 24 hours (denominator could be different if the recording period was actually <24 hours but ≥20 hours). Baseline assessment was based on 24-hour sound recordings using a digital recording device which recorded sounds from the lungs and trachea through a chest contact sensor, as well as ambient sounds through a lapel microphone. Population: All participants with 24-hour Coughs per Hour data available at baseline.
  coughs/hour
    number analyzed (Participants) | 232 | 235 | 237 | 704
    (all) | 38.07 (79.42) | 26.79 (21.13) | 28.53 (37.14) | 31.10 (52.04)

OUTCOME MEASURES:

1. Primary Outcome: Model-Based Geometric Mean Ratio (GMR) of 24-hour Objective Coughs Per Hour (Week 12/Baseline)
Description: 24-hour objective coughs per hour was defined as the total number of cough events during the monitoring period (24-hour interval) divided by 24 hours (denominator could be different if the recording period was actually <24 hours but ≥20 hours). Assessment was based on 24-hour sound recordings using a digital recording device which recorded sounds from the lungs and trachea through a chest contact sensor, as well as ambient sounds through a lapel microphone. A longitudinal analysis of covariance (ANCOVA) model was applied to log-transformed cough counts to determine geometric mean (GM) 24-hour objective coughs per hour at baseline and Week 12 on the original scale. The GMR corresponding to the Week 12 GM 24-hour objective coughs per hour divided by the Baseline GM 24-hour objective coughs per hour was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and provided at least 1 baseline and at least 1 Week 12 24-hour cough observation during the treatment period were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 222 | 227 | 217
ratio | 0.47 [0.41 to 0.54] | 0.48 [0.41 to 0.55] | 0.38 [0.33 to 0.44]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Estimated relative reduction (ERR) relative to Placebo (i.e. estimated percent change difference) was calculated by 100 (e**DIFF -1), where e = exponent of difference; and DIFF= treatment difference in change from baseline at Week 12 based on log transformed data; Test type: Other; p = 0.041, ANCOVA — Comparison based on a longitudinal ANCOVA model that included treatment, visit, treatment-by-visit interaction, gender, region, log-transformed baseline value, and log-transformed baseline value-by-visit as covariates; Estimated Percent Change Difference = -18.45, 95% CI 2-sided [-32.92 to -0.86]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.874, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Percent Change Difference = 1.56, 95% CI 2-sided [-16.13 to 22.99]

2. Primary Outcome: Number of Participants Experiencing At Least One Adverse Event (AE) During Treatment and Follow-up
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with at least one AE during either the 52-week treatment period or 2-week telephone follow-up was reported for all treatment study arms.
Time Frame: Up to approximately 54 weeks
Population: All randomized participants who received at least 1 dose of study intervention during the 52-week treatment period were analyzed. Per protocol, participants who continued in the optional Off-Treatment observational period were not included in the primary safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 243 | 244 | 243
Participants | 184 | 186 | 208

3. Primary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study intervention during the 52-week treatment period due to an AE for which the action taken was listed as 'drug withdrawn' was reported for all treatment study arms.
Time Frame: Up to approximately 52 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 243 | 244 | 243
Participants | 14 | 15 | 51

4. Secondary Outcome: Model-Based Geometric Mean Ratio (GMR) of Awake Objective Coughs Per Hour (Week 12/Baseline)
Description: Awake objective coughs per hour was defined as the total number of cough events during the monitoring period (24-hour interval) while the participant is awake divided by the total duration (in hours) for the monitoring period that the participant was awake. Assessment was based on 24-hour sound recordings using a digital recording device which recorded sounds from the lungs and trachea through a chest contact sensor, as well as ambient sounds through a lapel microphone. A longitudinal ANCOVA model was applied to log-transformed cough counts to determine GM awake objective coughs per hour at baseline and Week 12 on the original scale. The GMR corresponding to the Week 12 GM awake objective coughs per hour divided by the Baseline GM awake objective coughs per hour was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and provided at least 1 baseline and at least 1 Week 12 awake cough observation during the treatment period were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 222 | 227 | 217
ratio | 0.46 [0.40 to 0.53] | 0.47 [0.41 to 0.55] | 0.38 [0.33 to 0.44]
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.056, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Percent Change Difference = -17.68, 95% CI 2-sided [-32.57 to 0.50]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.770, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Estimated Percent Change Difference = 2.95, 95% CI 2-sided [-15.33 to 25.19]

5. Secondary Outcome: Percentage of Participants (Model-Based) With a ≤ -30% Change From Baseline in 24-hour Objective Coughs Per Hour at Week 12
Description: 24-hour coughs per hour was defined as the total number of cough events during the monitoring period (24-hour interval) divided by 24 hours (denominator could be different if the recording period was actually <24 hours but ≥20 hours). Assessment based on 24-hour sound recordings using a digital recording device. Percent change in 24-hour coughs per hour = (change from baseline in 24-hour coughs per hour / baseline 24-hour coughs per hour) ×100%. Negative values indicate a decrease in cough rate, while positive values indicate an increase in cough rate. A participant was considered a responder if the percent change from baseline in 24-hour coughs per hour was ≤ -30% (or a ≥30% reduction from baseline); a participant was considered a non-responder otherwise. The percentage of participants (logistic regression model-based) with a ≤ -30% change from baseline in 24-hour coughs per hour at Week 12 (≥30% reduction from baseline) was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and had available 24-hour cough data at baseline and at least one available post-baseline measurement were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 222 | 227 | 217
Percentage of Participants | 65.9 | 66.2 | 69.9
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline, and the interaction of baseline (underlying continuous response) by visit as covariates; Test type: Other; p = 0.416, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.77 to 1.86]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.948, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.66 to 1.55]

6. Secondary Outcome: Percentage of Participants (Model-Based) With a ≤ -1.3-point Change From Baseline in Mean Weekly Cough Severity Diary (CSD) Total Score at Week 12
Description: The CSD evaluates frequency of cough, intensity of cough and disruption and has a total of 7 items, each with scores ranging from 0 (best) to 10 (worst). The total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly total score was defined as the average of the mean total daily scores collected during the week prior to each visit. Baseline was defined as the average CSD scores collected during the week prior to Day 1 (Day -6 to Day 0). Participants were considered responders if the change from baseline in mean weekly CSD total score was ≤ -1.3 points (or a ≥1.3 point reduction from baseline); and considered a non-responder otherwise. Negative values indicate a decrease in cough severity, while positive values indicate an increase in cough severity. The percentage of participants (logistic regression model-based) with a ≤ -1.3 point change from baseline in CSD at Week 12 (or ≥1.3 point reduction from baseline) was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and had available CSD data at baseline and at least one available post-baseline measurement were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 237 | 241 | 234
Percentage of Participants | 52.4 | 62.1 | 60.5
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline CSD score, and the interaction of baseline (underlying continuous response) by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.94 to 2.05]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.01 to 2.18]

7. Secondary Outcome: Percentage of Participants (Model-Based) With a ≤ -2.7-point Change From Baseline in Mean Weekly CSD Total Score at Week 12
Description: The CSD evaluates frequency of cough, intensity of cough and disruption and has a total of 7 items, each with scores ranging from 0 (best) to 10 (worst). The total daily CSD score was the sum of these seven item scores (Min=0, Max=70). Mean weekly total score was defined as the average of the mean total daily scores collected during the week prior to each visit. Baseline was defined as the average CSD scores collected during the week prior to Day 1 (Day -6 to Day 0). Participants were considered responders if the change from baseline in mean weekly CSD total score was ≤ -2.7 points (or a ≥2.7 point reduction from baseline); and considered a non-responder otherwise. Negative values indicate a decrease in cough severity, while positive values indicate an increase in cough severity. The percentage of participants (logistic regression model-based) with a ≤ -2.7 point change from baseline in CSD at Week 12 (or ≥2.7 point reduction from baseline) was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 237 | 241 | 234
Percentage of Participants | 28.6 | 37.9 | 40.1
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.11 to 2.54]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.01 to 2.30]

8. Secondary Outcome: Percentage of Participants (Model-Based) With a ≤ -30 Millimeter (mm) Change From Baseline in Cough Severity Visual Analog Scale (VAS) Score at Week 12
Description: Cough severity was scored using the Cough Severity VAS, a single-item question asking the participant to rate the severity of their cough "today" using a 100 mm VAS (100-point scale) ranging from 0 ("No Cough") to 100 ("Extremely Severe Cough"). Mean weekly VAS score was derived as the average of VAS scores collected during the week prior to each visit. Baseline was defined as the average VAS scores collected during the week prior to Day 1 (Day -6 to Day 0). A participant was considered a responder if the change from baseline in mean weekly Cough Severity VAS score was ≤-30 mm (or a ≥30 mm reduction from baseline); participants considered non-responders otherwise. Negative values indicate a decrease in cough severity, while positive values indicate an increase in cough severity. The percentage of participants (logistic regression model-based) with ≤ -30 mm change from baseline in Cough Severity VAS at Week 12 (≥30 mm reduction from baseline) was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and had available Cough Severity VAS data at baseline and at least one available post-baseline measurement were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 237 | 241 | 234
Percentage of Participants | 31.3 | 36.7 | 41.2
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included treatment, visit, treatment-by-visit interaction, gender, region, baseline VAS score, and the interaction of baseline (underlying continuous response) by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.03 to 2.30]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 8, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.86 to 1.89]

9. Secondary Outcome: Percentage of Participants (Model-Based) With a ≥1.3-point Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score at Week 12
Description: The LCQ assesses the impact of chronic cough on health-related quality of life. It consists of 19 items which are divided over 3 domains: Physical (items 1, 2, 3, 9, 10, 11, 14 and 15), Psychological (4, 5, 6, 12, 13, 16, and 17), and Social (7, 8, 18, 19). A 7-point Likert scale is used to rate each item. For each domain, the domain score (range 1-7) is the sum of individual item score within the domain divided by the number of items in the domain. LCQ total score is the sum of the three domain scores and ranges from 3-21; with a higher score corresponding to a better health status. A participant was considered a responder if the change from baseline in LCQ total score was ≥1.3-points (increase from baseline); a participant was considered a non-responder otherwise. The percentage of participants (logistic regression model-based) with a ≥1.3-point change from baseline in LCQ total score at Week 12 was reported for all treatment study arms.
Time Frame: Baseline, Week 12
Population: All randomized participants in the analysis model who had taken at least 1 dose of study intervention and had available LCQ data at baseline and at least one available post-baseline measurement were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID
Number analyzed (Participants) | 217 | 226 | 214
Percentage of Participants | 61.3 | 68.8 | 67.3
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 45 mg BID; Comparison based on a logistic regression model that included visit, treatment-by-visit interaction, gender, region, baseline LCQ score, and the interaction of baseline (underlying continuous response) by visit as covariates; Test type: Other; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.85 to 1.98]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 15 mg BID; [analysis description as in outcome 9, analysis 1]; Test type: Other; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.92 to 2.12]

ADVERSE EVENTS:
Time Frame: On-Treatment Period (plus 2-week telephone follow-up): Up to Week 54; Off-Treatment (Off-Tx) Period: From Week 52 through Week 64 (approximately 12 weeks)
Description: All-Cause Mortality reported for all randomized participants by applicable treatment period. Serious and Other AEs include all randomized participants who received ≥1 dose of study drug during the Treatment Period. AEs were reported for a participant separately during the Treatment Period (MedDRA 23.0) and optional Off-Tx Period (MedDRA 23.1). Per protocol, only All-Cause Mortality, drug-related serious and nonserious AEs, and pregnancies were monitored during the Off-Tx Period.
Groups:
- Placebo: Off-Tx: Participants previously treated with dose-matched placebo BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
- Gefapixant 15 mg BID: Off-Tx: Participants previously treated with gefapixant 15 mg BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
- Gefapixant 45 mg BID: Off-Tx: Participants previously treated with gefapixant 45 mg BID for 52 weeks during the main study and extension study periods were observed for up to 3 months during an optional Off-Treatment Durability study period (participants received no treatment).
Arm/Group | Placebo | Gefapixant 15 mg BID | Gefapixant 45 mg BID | Placebo: Off-Tx | Gefapixant 15 mg BID: Off-Tx | Gefapixant 45 mg BID: Off-Tx
All-Cause Mortality (participants affected / at risk) | 2/244 | 1/244 | 0/244 | 0/10 | 0/18 | 0/13
Serious Adverse Events (participants affected / at risk) | 14/243 | 17/244 | 13/243 | 0/10 | 0/18 | 0/13
Other Adverse Events (participants affected / at risk) | 129/243 | 140/244 | 179/243 | 0/10 | 1/18 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=243) | Gefapixant 15 mg BID (N=244) | Gefapixant 45 mg BID (N=243) | Placebo: Off-Tx (N=10) | Gefapixant 15 mg BID: Off-Tx (N=18) | Gefapixant 45 mg BID: Off-Tx (N=13)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilloma viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=243) | Gefapixant 15 mg BID (N=244) | Gefapixant 45 mg BID (N=243) | Placebo: Off-Tx (N=10) | Gefapixant 15 mg BID: Off-Tx (N=18) | Gefapixant 45 mg BID: Off-Tx (N=13)
Diarrhoea (Gastrointestinal disorders) | 14 (19) | 15 (19) | 12 (23) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 7 (7) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (22) | 8 (8) | 17 (20) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 11 (12) | 20 (25) | 11 (17) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 51 (75) | 47 (60) | 50 (63) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 18 (20) | 13 (19) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (14) | 14 (14) | 9 (13) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 13 (18) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 14 (17) | 20 (27) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 3 (5) | 33 (37) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 8 (9) | 22 (25) | 88 (101) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 31 (55) | 34 (57) | 29 (51) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 5 (5) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 2 (2) | 24 (24) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 9 (10) | 11 (18) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 14 (14) | 16 (17) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 13 (18) | 14 (14) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission to allow the Sponsor to protect proprietary information and comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03449134/Prot_SAP_000.pdf